CLINICAL TRIAL: NCT01662986
Title: A Randomized, Placebo-controlled, Double-blind, Parallel Group, Multi Center Study to Assess the Safety and Efficacy of Tiotropium Bromide (18 µg) Delivered Via the HandiHaler® in Chronic Obstructive Pulmonary Disease (COPD) Subjects Recovering From Hospitalization for an Acute Exacerbation (Hospital Discharge Study 2)
Brief Title: Investigate the Impact of Early Treatment Initiation With Tiotropium in Patients Recovering From Hospitalization for an Acute COPD Exacerbation 2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.478
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Results first posted 2015-07-20 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

ARMS (2):
- 18 mcg tiotropium bromide (Active Comparator): Patient to receive one tiotropium bromide inhalation powder capsule daily (in the morning) via HandiHaler
  Interventions: Drug: tiotropium bromide
- placebo (Placebo Comparator): Patient to receive one placebo inhalation powder capsule daily (in the morning) via HandiHaler
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tiotropium bromide — 18 mcg once a day (QD)
  Arms: 18 mcg tiotropium bromide
Drug: Placebo — Once a day (QD)
  Arms: placebo

SUMMARY:
A randomized, placebo-controlled, double-blind, parallel group, multi-center study to assess the safety and efficacy of tiotropium bromide (18 µg) delivered via the HandiHaler® in Chronic Obstructive Pulmonary Disease (COPD) subjects recovering from hospitalization for an acute exacerbation (Hospital Discharge Study 2)

ELIGIBILITY:
Inclusion criteria:

The following inclusion criteria apply at Visit 0:

1. All subjects must sign an informed consent consistent with the International Conference on Harmonization - Good Clinical Practice (ICH-GCP) guidelines prior to participation in the trial and conducting any study procedures
2. Male or female subjects 40 years of age or older.
3. Hospitalization for a primary diagnosis of acute COPD exacerbation for =14 days. Determination of accuracy of admission diagnosis will be at the discretion of the investigator.
4. Patient reported hospital length of stay and discharge date (confirmed with hospital discharge summary/hospital records; however, medical record confirmation may occur following randomization).

   The following inclusion criteria apply at Visit 1:
5. Discharged from the hospital =10 days from date of randomization.
6. All subjects must have a diagnosis of COPD (P12-01205), and have documented airway obstruction with a post-bronchodilator Force Expiratory Volume in 1 second (FEV1)\ Force vital capacity (FVC) <0.7(See Section 5.1.2, Pulmonary Function Testing). The diagnosis of COPD can be made at Visit 1 if no Pulmonary Function Testing (PFT) data available within the past 12 months.
7. Subjects must be current or ex-smoker with a smoking history of =10 pack-years:

Pack-years = Number of cigarettes/day x years of smoking 20 cigarettes/ pack 8. Subjects must be able to inhale medication in a competent manner from the HandiHaler® device (Appendix 10.1) and from a metered dose inhaler (MDI).

Exclusion criteria:

The following exclusion criterion applies at Visit 0:

1. No more than 30 days of therapy with any long-acting inhaled anticholinergic over preceding 3 months prior to discharge from the hospital, and no therapy with any long acting anticholinergic post discharge (no use between hospital discharge and randomization) or any other restricted concomitant medications

   The following exclusion criteria apply at Visit 1:
2. Presence of a significant disease (in the opinion of the investigator) which may put the subject at risk because of participation in the study or may influence the subject's ability to participate in the study for up to 2 years.
3. A documented history of myocardial infarction during the hospitalization preceding randomization. Subjects being stable with a history of cardiac stents are permitted.
4. Any unstable or life-threatening cardiac arrhythmia requiring intervention or change in drug therapy during the last year.
5. Subjects with asthma (subject treated for asthma in the last 2 years, history of childhood asthma is permitted), cystic fibrosis, clinical diagnosis of bronchiectasis, interstitial lung disease, pulmonary thromboembolic disease or known active tuberculosis.

7. Malignancy for which the subject has undergone resection, radiation, chemotherapy or biological treatments within the last two years or is currently on active radiation therapy, chemotherapy or biological treatment. Subjects with treated basal cell carcinoma and non-invasive squamous cell skin carcinoma are allowed.

8. Hospitalization for cardiac failure (New York Heart Association (NYHA) class III or IV) during the hospitalization preceding randomization.

9. Known hypersensitivity to anticholinergic drugs, lactose, or any other components of the HandiHaler® or MDI inhalation solution delivery system.

10. Known moderate to severe renal impairment as judged by the investigator. 11. Known narrow angle glaucoma as judged by the investigator. 12. Significant symptomatic prostatic hyperplasia or bladder-neck obstruction. Subjects whose symptoms are controlled on treatment may be included.

13. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (i.e., oral contraceptives, intrauterine devices, diaphragm or sub dermal implants e.g., Norplant®) for at least three months prior to and for the duration of the trial.

14. Significant alcohol or drug abuse within the past 12 months. 15. Previously randomized in this study or currently participating in another interventional study.

16. Visual impairment that as judged by the investigator does not allow the subject to independently read and complete the questionnaires and eDiary.

17. Any significant or new ECG findings at Visit 1 as judged by the investigator, including, but not limited to signs of acute ischemia, arrhythmia.

18. Treatment with any restricted pulmonary medication. 19. Residing in an assisted living facility.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2014-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (50):
- United States (50):
  - 205.478.00243 Boehringer Ingelheim Investigational Site, Montgomery, Alabama
  - 205.478.00208 Boehringer Ingelheim Investigational Site, Flagstaff, Arizona
  - 205.478.00260 Boehringer Ingelheim Investigational Site, Glendale, Arizona
  - 205.478.00241 Boehringer Ingelheim Investigational Site, Loma Linda, California
  - 205.478.00240 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 205.478.00237 Boehringer Ingelheim Investigational Site, Torrance, California
  - 205.478.00231 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 205.478.00209 Boehringer Ingelheim Investigational Site, Danbury, Connecticut
  - 205.478.00250 Boehringer Ingelheim Investigational Site, Glastonbury, Connecticut
  - 205.478.00229 Boehringer Ingelheim Investigational Site, Hartford, Connecticut
  - 205.478.00200 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 205.478.00212 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 205.478.00265 Boehringer Ingelheim Investigational Site, Kissimmee, Florida
  - 205.478.00246 Boehringer Ingelheim Investigational Site, Lehigh Acres, Florida
  - 205.478.00248 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 205.478.00215 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 205.478.00261 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 205.478.00233 Boehringer Ingelheim Investigational Site, Vero Beach, Florida
  - 205.478.00236 Boehringer Ingelheim Investigational Site, Austell, Georgia
  - 205.478.00205 Boehringer Ingelheim Investigational Site, Lawrenceville, Georgia
  - 205.478.00225 Boehringer Ingelheim Investigational Site, Evanston, Illinois
  - 205.478.00264 Boehringer Ingelheim Investigational Site, Iowa City, Iowa
  - 205.478.00254 Boehringer Ingelheim Investigational Site, Olathe, Kansas
  - 205.478.00249 Boehringer Ingelheim Investigational Site, Topeka, Kansas
  - 205.478.00257 Boehringer Ingelheim Investigational Site, Hazard, Kentucky
  - 205.478.00234 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 205.478.00242 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 205.478.00258 Boehringer Ingelheim Investigational Site, Eunice, Louisiana
  - 205.478.00256 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 205.478.00210 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 205.478.00220 Boehringer Ingelheim Investigational Site, Towson, Maryland
  - 205.478.00204 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 205.478.00247 Boehringer Ingelheim Investigational Site, Winston Salem, Massachusetts
  - 205.478.00263 Boehringer Ingelheim Investigational Site, Rochester, Minnesota
  - 205.478.00201 Boehringer Ingelheim Investigational Site, Chesterfield, Missouri
  - 205.478.00239 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 205.478.00227 Boehringer Ingelheim Investigational Site, Summit, New Jersey
  - 205.478.00253 Boehringer Ingelheim Investigational Site, The Bronx, New York
  - 205.478.00226 Boehringer Ingelheim Investigational Site, Chapel Hill, North Carolina
  - 205.478.00232 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 205.478.00203 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 205.478.00206 Boehringer Ingelheim Investigational Site, Wyomissing, Pennsylvania
  - 205.478.00219 Boehringer Ingelheim Investigational Site, Easley, South Carolina
  - 205.478.00222 Boehringer Ingelheim Investigational Site, Arlington, Texas
  - 205.478.00235 Boehringer Ingelheim Investigational Site, Kingwood, Texas
  - 205.478.00217 Boehringer Ingelheim Investigational Site, McKinney, Texas
  - 205.478.00216 Boehringer Ingelheim Investigational Site, Temple, Texas
  - 205.478.00230 Boehringer Ingelheim Investigational Site, Falls Church, Virginia
  - 205.478.00202 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 205.478.00224 Boehringer Ingelheim Investigational Site, Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomized, placebo-controlled, double blind, parallel group design involving an event-driven treatment period up to the close of the study and a minimum 30-day follow-up period up to the close of the study
Groups:
- Placebo: Patient to receive oral inhalation of one placebo powder capsule once daily in the morning via HandiHaler.
- Tiotropium Bromide (18 μg): Patient to receive oral inhalation of one tiotropium bromide powder capsule once daily in the morning via HandiHaler
Period: Overall Study
Arm/Group | Placebo | Tiotropium Bromide (18 μg)
Started | 40 | 39
Completed | 22 | 26
Not Completed | 18 | 13
Not completed — Adverse Event | 5 | 4
Not completed — Protocol Violation | 2 | 3
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Not Treated | 1 | 0
Not completed — Other than stated above | 3 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all patients randomized and who took at least one dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tiotropium Bromide (18 μg) | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.0 (8.6) | 58.4 (7.0) | 59.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Trough FEV1 at 12 Weeks on Study Drug.
Description: Change from baseline of trough forced expiratory volume in 1 second (FEV1) at 12 weeks on study drug.
  Trough FEV1 is defined as the FEV1 measurement prior to the next dosing of study drug and approximately 24 hours after last inhalation of drug.
Time Frame: Baseline and 12 weeks
Population: Treated Set (TS): The treated set included all patients randomized and who took at least one dose of the study drug. The number of patients analyzed at week 12 from the treated set were 29 for Placebo and 30 for Tiotropium.
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Placebo | Tiotropium Bromide (18 μg)
Number analyzed (Participants) | 29 | 30
Litres | 0.124 (0.271) | 0.186 (0.475)

2. Secondary Outcome: Change From Baseline of Trough FVC at 12 Weeks on Study Drug.
Description: Change from baseline of trough Forced Vital Capacity (FVC) at 12 weeks on study drug.
Time Frame: baseline and 12 weeks
Population: Treated Set (TS). The number of patients analyzed at week 12 from the treated set were 29 for Placebo and 30 for Tiotropium.
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Placebo | Tiotropium Bromide (18 μg)
Number analyzed (Participants) | 29 | 30
Litres | 0.090 (0.399) | 0.282 (0.558)

3. Secondary Outcome: Percentage of Patients With Adverse Clinical Event During on Study.
Description: Percentage (number) of patients with adverse clinical event on study, which is defined as the combined endpoint of Chronic obstructive pulmonary disease (COPD) exacerbations per Boehringer Ingelheim (BI) definition, all-cause re-hospitalization, or all-cause mortality.
Time Frame: from first drug administration to the last timepoint with information of clinical adverse outcome available, Up to 2 years
Population: Treated Set (TS)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tiotropium Bromide (18 μg)
Number analyzed (Participants) | 39 | 39
percentage of participants | 35.9 | 46.2

4. Secondary Outcome: Change From Baseline of Trough FEV1 at 12 Weeks on Study Drug From the Two Twin Trials, Present 205.478 (NCT01662986) and 205.477 (NCT01663987)
Description: Change from baseline of trough FEV1 (forced expiratory volume in 1 second) at 12 weeks on study drug.
  Trough FEV1 is defined as the FEV1 measurement prior to the next dosing of study drug and approximately 24 hours after last inhalation of drug.
Time Frame: Baseline and week 12
Population: Treated Set of the pooled twin studies 205.478 and 205.477. The number of patients analyzed at week 12 from the treated set were 59 for Placebo and 60 for Tiotropium.
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Placebo | Tiotropium Bromide (18 μg)
Number analyzed (Participants) | 59 | 60
Litres | 0.035 (0.262) | 0.185 (0.384)

5. Secondary Outcome: Change From Baseline of Trough FVC at 12 Weeks From the Two Twin Trials, Present 205.478 (NCT01662986) and 205.477 (NCT01663987)
Description: Change from baseline of trough Forced Vital Capacity (FVC) at 12 weeks on study drug.
Time Frame: Baseline and week 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Placebo | Tiotropium Bromide (18 μg)
Number analyzed (Participants) | 59 | 60
Litres | -0.015 (0.396) | 0.278 (0.447)

6. Secondary Outcome: Percentage of Patients With COPD Exacerbation From the Two Twin Trials, Present 205.478 (NCT01662986) and 205.477 (NCT01663987)
Description: Percentage (number) of patients with COPD exacerbation on study was analysed for the combined study.
  A COPD exacerbation was defined as a complex of lower respiratory events/symptoms (increase or new onset) related to the underlying COPD with duration of three days or more, requiring a change in treatment where a complex of lower respiratory events/symptoms was defined as at least two of the following:
  1) Shortness of breath; 2) Sputum production (volume) ; 3) Occurrence of purulent sputum; 4) Cough; 5) Wheezing; 6) Chest tightness.
  Onset of exacerbation was defined by the onset of first recorded symptom.The end of exacerbation was decided by the investigator based on clinical judgment.
  A required change in treatment included either prescription of antibiotics and/or systemic steroids; and/or a newly prescribed maintenance respiratory medication (i.e., bronchodilators including theophyllines and PDE4-inhibitors).
Time Frame: as for outcome 3
Population: Treated Set of the pooled twin studies 205.478 and 205.477
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tiotropium Bromide (18 μg)
Number analyzed (Participants) | 78 | 79
percentage of participants | 44.9 | 40.5

7. Secondary Outcome: Percentage of Patients With All-cause Hospitalization From the Two Twin Trials, Present 205.478 (NCT01662986) and 205.477 (NCT01663987).
Description: Percentage (number) of patients with all-cause hospitalization outcome event occured during the study was analysed for the combined study.
  All-cause hospitalization included all hospitalizations, except planned hospitalizations for elective procedures.
  Hospitalizations occurring on the same day as discharge were not considered a separate admission.
Time Frame: as for outcome 3
Population: Treated Set of the pooled twin studies 205.478 and 205.477
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tiotropium Bromide (18 μg)
Number analyzed (Participants) | 78 | 79
percentage of participants | 26.9 | 26.6

8. Secondary Outcome: Percentage of Patients With 30-day Hospital Readmission Rates Outcome Event From the Two Twin Trials, Present 205.478 (NCT01662986) and 205.477 (NCT01663987)
Description: Percentage (number) of patients with 30-day hospital readmission rates outcome events was analysed.
  Days to hospital readmission were calculated as:Hospital readmission days = Readmission date - Date of hospital discharge + 1.
  The 30-day hospital readmission analysis summarized the frequency of patients with hospital readmission and readmission days >1 and <31 days using the TS.
Time Frame: from date of hospital discharge prior to randomization upto readmission days >1 and <31 days
Population: Treated Set of the pooled twin studies 205.478 and 205.477
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tiotropium Bromide (18 μg)
Number analyzed (Participants) | 78 | 79
percentage of participants | 5.1 | 5.1

9. Secondary Outcome: Number of COPD Exacerbation Events From the Two Twin Trials, Present 205.478 (NCT01662986) and 205.477 (NCT01663987)
Description: Number of COPD exacerbation per patient year outcome event occured during the study was analysed descriptively by calculating average occurrence (number of events per patient year drug exposure) by treatment group for on study period using the TS.
Time Frame: start of treatment to the last timepoint with information of clinical adverse outcome available,Up to 2 years
Population: Treated Set of the pooled twin studies 205.478 and 205.477. The number of patients analyzed for this endpoint from the treated set were 73 for Placebo and 54 for Tiotropium.
Measure: Number; unit: exacerbations per patient year
Arm/Group | Placebo | Tiotropium Bromide (18 μg)
Number analyzed (Participants) | 73 | 54
exacerbations per patient year | 1.3 | 0.9

10. Secondary Outcome: Exposure of COPD Exacerbation Events From the Two Twin Trials, Present 205.478 (NCT01662986) and 205.477 (NCT01663987)
Description: Total patient year exposure of COPD was calculated by aggregating the time to min(treatment stop +30, last contact) for on-treatment analysis, or time to last contact for on-study analysis.
Time Frame: start of treatment to the last timepoint with information of clinical adverse outcome available,Up to 2 years
Population: as for outcome 9
Measure: Number; unit: Patient years
Arm/Group | Placebo | Tiotropium Bromide (18 μg)
Number analyzed (Participants) | 73 | 54
Patient years | 58.0 | 60.2

11. Primary Outcome: Percentage of Patients With Next Adverse Clinical Outcome Event From the Two Twin Trials, Present 205.478 (NCT01662986) and 205.477 (NCT01663987).
Description: Percentage (number) of patients with next adverse clinical outcome event occured during the study, defined as the combined endpoint of Chronic obstructive pulmonary disease (COPD) exacerbations per Boehringer Ingelheim (BI) definition, all-cause re-hospitalization, or all-cause mortality.
  Time to the next adverse clinical outcome event from the Two Twin Trials, present 205.478 (NCT01662986) and 205.477 (NCT01663987) was not analysed, only Kaplan Meier curve was plotted. So this endpoint has not been disclosed.
  This endpoint was analysed using combined data, as specified in the analysis plan
Time Frame: as for outcome 3
Population: Treated Set of the pooled twin studies 205.478 and 205.477 : This set includes all patients who were randomized and took at least one dose of the study drug, 157 patients (79 tiotropium and 78 placebo) were included in this set.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Tiotropium Bromide (18 μg)
Number analyzed (Participants) | 78 | 79
Percentage of participants | 47.4 | 53.2

12. Secondary Outcome: Number of All-cause Hospitalization Event From the Two Twin Trials, Present 205.478 (NCT01662986) and 205.477 (NCT01663987)
Description: Number of all-cause hospitalization per patient year outcome event occured during the study was analysed descriptively by calculating average occurrence (number of events per patient year drug exposure) by treatment group for on study period using the TS.
Time Frame: as for outcome 3
Population: Treated Set of the pooled twin studies 205.478 and 205.477. The number of patients analyzed for this endpoint from the treated set were 47 for Placebo and 38 for Tiotropium.
Measure: Number; unit: hospitalizations per patient year
Arm/Group | Placebo | Tiotropium Bromide (18 μg)
Number analyzed (Participants) | 47 | 38
hospitalizations per patient year | 0.8 | 0.6

13. Secondary Outcome: Exposure of All-cause Hospitalization Event From the Two Twin Trials, Present 205.478 (NCT01662986) and 205.477 (NCT01663987)
Description: Total patient year exposure of all-cause hospitalization was calculated by aggregating the time to min(treatment stop +30, last contact) for on-treatment analysis, or time to last contact for on-study analysis.
Time Frame: as for outcome 3
Population: as for outcome 12
Measure: Number; unit: patient years
Arm/Group | Placebo | Tiotropium Bromide (18 μg)
Number analyzed (Participants) | 47 | 38
patient years | 58.0 | 60.2

14. Secondary Outcome: Time to Event: Time to Recovery (EXACT-PRO) From the Two Twin Trials, Present 205.478 (NCT01662986) and 205.477 (NCT01663987)
Description: Time to event: Time to recovery based on EXACT-PRO total score. The percentage of observed patients recovered by end of study was reported.
  Time to recovery was assessed with the EXACT-PRO questionnaire. EXACT-PRO total scores were transformed to smooth scores for determining time to recovery and all other endpoints related to the EXACT questionnaire. The day-2 score was transformed to the mean of the total scores recorded on Day 1, 2, and 3. Similarly, each subsequent day's score was transformed to the mean score using a rolling 3-day average.
  Analysis based on Kaplan Meier estimate
Time Frame: from first drug administration to the last timepoint with information of EXACT-PRO, Up to 2 years
Population: Patients who had baseline and post-baseline measurements of EXACT-PRO.
Measure: Number; unit: Percentage of patients recovered
Arm/Group | Placebo | Tiotropium Bromide (18 μg)
Number analyzed (Participants) | 76 | 76
Percentage of patients recovered | 94.0 | 88.0

ADVERSE EVENTS:
Time Frame: From first drug administration until 30 days after the last drug administration, up to 405 days
Groups:
- Placebo: Patient to receive one placebo inhalation powder capsule once daily in the morning via HandiHaler
Arm/Group | Placebo | Tiotropium Bromide (18 μg)
Serious Adverse Events (participants affected / at risk) | 9/39 | 10/39
Other Adverse Events (participants affected / at risk) | 11/39 | 23/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=39) | Tiotropium Bromide (18 μg) (N=39)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Substance abuse (Psychiatric disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=39) | Tiotropium Bromide (18 μg) (N=39)
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Chest discomfort (General disorders) | 0 | 2
Chest pain (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 0 | 3
Bronchitis (Infections and infestations) | 1 | 2
Candida infection (Infections and infestations) | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
The original protocol planned to randomize 604 subjects. However this was not reached due to low patient enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.